CLINICAL TRIAL: NCT00738244
Title: Methods of Wind Noise Suppression in Hearing Aids
Brief Title: Effectiveness of Hearing-aid Based Wind-noise Algorithm
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Ruth Ann Bentler, Professor, University of Iowa
Other Study IDs: 2R44DC007246-02A2 (NIH); R44DC007246 (NIH)
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Hearing Impairment
Keywords: hearing aid algorithm; wind-noise suppression
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Normal hearing listeners
- 2: Listeners with mild-to-moderate sensorineural hearing loss

SUMMARY:
Wind-noise is highly disturbing to hearing impaired individuals wearing hearing aids who wish to participate in outdoor conversations where wind is present or during activities such as walking or running. In these situations, wind noise significantly reduces signal-to-noise ratio and, consequently, the intelligibility of speech and sounds may be significantly impaired. This negative effect is exacerbated with the use of directional microphone schemes in the hearing iads. The objective of this project is to determine the efficacy of the MH Acoustics' multi-microphone wind-noise reduction invention for the digital hearing aids market. MH Acoustics' wind noise reduction technology is unique since it provides instantaneous convergence while maintaining directionality of the microphone array. Current commercial technologies do not provide this feature. We are hypothesizing that, due to the design of the algorithm, speech perception ability and sound quality perception will be better than that available with traditional directional and/or omnidirectional microphone schemes in windy environments.

DETAILED DESCRIPTION:
Two groups of subjects will be recruited to participate: Normal hearing adults and adults with mild to moderately severe hearing loss, ages 18-65. Pure tone audiometrics (re ANSI, 1996) will be done to ascertain the hearing sensitivity through 6ooo Hz. Normal hearing will be defined as thresholds at or better than 20 dB HL (re ANSI, 1996). The only exclusion criterion for the group exhibiting hearing loss is that no thresholds up to and including 3000 Hz will exceed 75 dB, so as to minimize the inclusion of subjects with "dead regions" in the cochlea.

Subjects will be seen for four visits to the laboratory. The first visit will involve documentation of informed consent, and measurement of hearing thresholds. The second, third and fourth visits will consist of testing with the following measures (in random order for each subject) to determine if the various implementations of the wind noise reduction algorithm 1) impact speech perception ability, and/or 2) impact sound quality perception. Each session will take approximately 1.5 hours, with a maximum of six hours over all the sessions. The two speech perception tests that will be utilized include : 1) Connected Speech Test and Hearing in Noise Test, 2) The Hearing in Noise Test (HINT) (Nilsson, Soli, & Sullivan, 1994; Koch, Nilsson & Soli, 1995. Overall Impression of Sound Quality and Ratings of Annoyance will be used as subjective, or self-reported, measures of preference. Overall Impression will be influenced by the audibility and masking effect of the noise bursts, whereas Annoyance ratings are significantly correlated to the high frequency emphasis of the stimulus, a potential impact of the extreme suppression conditions (e.g., -18 dB) (Warner & Bentler, 2002; Miedema & Vos, 2003). Both measures will be analyzed as a function of the different time constants, gain reduction levels, and level of presentation.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-75
* Normal or mild-to-moderate sensorineural hearing loss

Exclusion Criteria:

* Thresholds in excess of 75 dB HL

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups (30 each) of subjects will be recruited to participate: Normal hearing adults and adults with mild to moderately severe hearing loss, ages 18-65. Pure tone audiometrics (re ANSI, 1996) will be done to ascertain the hearing sensitivity through 6ooo Hz. Normal hearing will be defined as thresholds at or better than 20 dB HL (re ANSI, 1996). The only exclusion criterion for the group exhibiting hearing loss is that no thresholds up to and including 3000 Hz will exceed 75 dB, so as to minimize the inclusion of subjects with "dead regions" in the cochlea.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Speech Perception as measured by the Connected Speech Test (Cox et al) | Each of three follow-up visits

SECONDARY OUTCOMES:
Sound Quality | Each of three follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A Bentler, PhD, Principal Investigator — University of Iowa
Locations (1):
- Wendell Johnson Center, University of Iowa, Iowa City, Iowa, United States